CLINICAL TRIAL: NCT00715650
Title: Benefits Counseling to Preserve Function Among Disability Applicants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D6432-R
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Veterans' Disability Claims
Keywords: Rehabilitation, Vocational; Compensation and Redress; disability evaluation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): This counseling consists of four sessions each approximately 60 minutes each. The four sessions are organized as follows: a) Orientation to Benefits Counseling: Your Benefits and Your Goals b) Work and Claims c) Financial Review: Implications of Your Work Plan and d) Your Plans After the Benefits Notice. The first session focuses on the disability application process as a non-confrontational way to explore attitudes towards work. The second session more directly addresses the claimant's attitudes about work and beliefs about whether work will prevent receipt of disability benefits. The third session addresses the same issue as the second, ambivalence about work and disability, from a financial perspective. The fourth session occurs after the disability determination has been made, and it is possible the veteran may feel differently about a benefit that has been awarded.
  Interventions: Behavioral: Benefits Counseling
- Arm 2 (Active Comparator): This will consist of four-session orientation with the sessions organized as follows: a) overview of VHA services, b) Primary Care c) Pharmacy and laboratory services and d) specialty services. After the description of each service, participants will be invited to discuss which services they plan to utilize. The counselor will provide telephone numbers and directions to the sites at which these services are provided.
  Interventions: Behavioral: VA Orientation

INTERVENTIONS:
Behavioral: Benefits Counseling — Benefits counseling is designed to improve the quality of life of disability applicants by accomplishing two functions: 1) Providing information concerning what vocational rehabilitation services are available and how they will affect receipt of disability payments, 2) Amplifying applicants' existing motivation to engage in work and related-activities, using a Motivational Interviewing approach.
  Other Names: Motivational Interviewing
  Arms: Arm 1
Behavioral: VA Orientation — VA Orientation is designed to provide the Veteran with information regarding the services available, how to access the services and where the service is located on the VA campus.
  Other Names: New patient orientation
  Arms: Arm 2

SUMMARY:
This study will address the problem that claimants with psychiatric disabilities who apply for and receive disability benefits go on to work less than those whose claims are denied.

DETAILED DESCRIPTION:
The objective of this research is to conduct a 6-month randomized clinical trial comparing participants assigned to Benefits Counseling and to those assigned to the control condition, VA Orientation. Benefits Counseling is an adaptation of two counseling approaches to foster veterans' involvement in work and work-related activity compared to the control condition, VA Orientation. The first approach helped recipients of Social Security disability benefits for psychiatric illness return to work in part by alleviating beneficiaries' concerns that they would lose their benefits if they worked. The second approach is a Motivational Interviewing approach that showed great promise in engaging veterans with psychiatric disabilities in compensated work therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has never received VBA benefits
* Able to provide valid consent
* Expresses willingness to discuss benefits with a counselor
* Difficulty working as evidenced by a "Yes" to either (a), (b), or (c) of the question below about work-related difficulties: During the past 4 weeks, have you had any of the following problems (such as feeling depressed and anxious):

  * Cut down on the amount of time you spent on work or other activities?
  * Accomplished less than you would like?
  * Didn't do work or other activities as carefully as usual?
* Expresses willingness to try Benefits Counseling if assigned to it
* An evaluation by a psychiatrist or psychologist is scheduled

Exclusion Criteria:

* Already receiving VA payments
* Already receiving SSI or SSDI payments
* Has a conservator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

REFERENCES:
- [Result] Meshberg-Cohen S, Reid-Quinones K, Black AC, Rosen MI. Veterans' attitudes toward work and disability compensation: associations with substance abuse. Addict Behav. 2014 Feb;39(2):445-8. doi: 10.1016/j.addbeh.2013.09.005. Epub 2013 Sep 11. PMID 24090622
- [Result] Rosen MI, Ablondi K, Black AC, Mueller L, Serowik KL, Martino S, Mobo BH, Rosenheck RA. Work outcomes after benefits counseling among veterans applying for service connection for a psychiatric condition. Psychiatr Serv. 2014 Dec 1;65(12):1426-32. doi: 10.1176/appi.ps.201300478. Epub 2014 Oct 31. PMID 25082304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from December 2008 to December 2011. Veterans were eligible for participation if they were seeking service-connection for a psychiatric disability and they indicated that emotional problems had interfered with work in the past 28 days.
Groups:
- Benefits Counseling: Four 50-minutes sessions of individual counseling using motivational interviewing to increase veterans' desire to engage in work and related activities
- VA Orientation: Four sessions of VA orientation that taught veterans about the VA health care system generally and about the specific general medical and mental health services available to veterans
Period: Intervention
Arm/Group | Benefits Counseling | VA Orientation
Started | 47 | 45
Received Any Session | 39 | 38
Attended ≥ 2 Sessions | 36 | 33
Attended ≥ 3 Sessions | 23 | 17
Completed | 42 | 42
Not Completed | 5 | 3
Period: Follow-up
Arm/Group | Benefits Counseling | VA Orientation
Started | 42 | 42
Completed Month 1 Follow-up | 40 | 38
Completed Month 3 Follow-up | 35 | 40
Completed Month 6 Follow-up | 29 | 37
Completed | 29 | 37
Not Completed | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benefits Counseling | VA Orientation | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (4) | 40 (14) | 38.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 32 | 38 | 70
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 28 | 53
  African American | 6 | 5 | 11
  Latino | 8 | 5 | 13
  Other | 3 | 4 | 7
Psychiatric diagnosis [Number; unit: participants]
  Major depression | 15 | 10 | 25
  PTSD | 9 | 15 | 24
  TBI | 1 | 3 | 4
  Schizophrenia type/Bipolar | 3 | 2 | 5
  Substance abuse | 11 | 6 | 17
Attitudes and beliefs: "If a person is receiving VA benefits and starts working for pay ..." [Mean (Standard Deviation); unit: Likert scale] — Veterans were asked to rate their agreement with three statements asserting a relationship between work and receipt of disability payments. Agreement was rated on a 4-point, forced-choice Likert scale anchored by strongly disagree (1), somewhat disagree (2), somewhat agree (3), and strongly agree (4).
  Likert scale
    Income benefits will be reduced or stopped | 3.4 (1.4) | 3.5 (1.2) | 3.45 (1.4)
    Medical benefits will remain the same | 3.1 (1.4) | 2.8 (1.3) | 2.95 (1.4)
    Would rather turn down job than lose benefits | 3.3 (1.0) | 3.6 (1.0) | 3.45 (1)

OUTCOME MEASURES:

1. Primary Outcome: Days of Work and Work-related Activity
Description: Number of days in the past 28 spent engaged in any kind of work or related activity. Measured using a timeline follow-back calendar.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benefits Counseling | VA Orientation
Number analyzed (Participants) | 42 | 42
days
  Any work activity | 8.3 (8.1) | 8.7 (9.4)
  Work for pay | 6.6 (8.8) | 9.0 (10.1)
  Work for no pay | .3 (1.2) | .1 (.2)
  Classes | 2.6 (6.2) | 1.6 (4.9)
  Vocational rehabilitation | .1 (.3) | .0 (.2)

2. Primary Outcome: Days of Work and Work-related Activity
Description: as for outcome 1
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benefits Counseling | VA Orientation
Number analyzed (Participants) | 42 | 42
days
  Any work activity | 8.6 (9.1) | 9.8 (10.0)
  Work for pay | 7.0 (9.3) | 10.0 (10.3)
  Work for no pay | 1.4 (1.7) | 3.3 (.5)
  Classes | 3.7 (3.7) | 4.6 (1.0)
  Vocational rehabilitation | 4.5 (.4) | 0 (.4)

3. Primary Outcome: Days of Work and Work-related Activity
Description: as for outcome 1
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benefits Counseling | VA Orientation
Number analyzed (Participants) | 42 | 42
days
  Any work activity | 11.6 (8.9) | 11.6 (9.5)
  Work for pay | 9.3 (9.3) | 10.3 (10.3)
  Work for no pay | 1.7 (5.2) | .5 (2.1)
  Classes | 3.7 (7.0) | 1.0 (3.1)
  Vocational rehabilitation | .4 (2.1) | .4 (2.5)

4. Primary Outcome: Days of Work and Work-related Activity
Description: as for outcome 1
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benefits Counseling | VA Orientation
Number analyzed (Participants) | 42 | 42
days
  Any work activity | 12.7 (8.4) | 10.5 (9.4)
  Work for pay | 10.5 (9.6) | 7.8 (9.6)
  Work for no pay | 2.6 (6.1) | 1.4 (4.7)
  Classes | 4.8 (8.5) | 2.5 (5.9)
  Vocational rehabilitation | .6 (3.0) | .3 (1.7)

ADVERSE EVENTS:
Arm/Group | Benefits Counseling | VA Orientation
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No